CLINICAL TRIAL: NCT03431116
Title: The Prediction of Risk Factors of Progression of Low Implanted Placenta at 18- 24 Weeks to Placenta Previa at Term
Brief Title: Low Implanted Second Trimester Placenta and Placenta Previa
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Other Study IDs: PPLIP
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low implanted placenta group
  Interventions: Radiation: ultrasound

INTERVENTIONS:
Radiation: ultrasound — to detect the placental site

SUMMARY:
Placenta Previa is defined as a placenta implanted in the lower segment of the uterus, presenting ahead of the leading pole of the fetus (over or near the internal os). The prevalence of placenta previa has been estimated to be approximately 0.5% of all pregnancies, and this increase correlates to the elevated cesarean section rate . In Egypt, the prevalence of placenta previa is around 1.3% in Sohag Governorate and 1.5% in Aswan region according to.

Although various studies have tried to address risk factors associated with Placenta Previa development, the etiology of placenta previa still remains obscure. Several risk actors have been identified as strong contributors to placenta previa development. It is also a significant contributor to severe postpartum hemorrhage.Risk factors include; history of previous cesarean section, advanced maternal age, history of previous abortions, high parity and substance abuse during pregnancy (cigarette smoking), placental size (multiple pregnancy), endometrial damage (previous dilatation and curettage), uterine scars and pathology (previous myomectomy or endometritis), placental pathology (marginal cord insertions and succenturiate lobes), previous placental Previa, and curiously.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 18-24 weeks.
2. Diagnosed to have low implanted placenta by ultrasound

Exclusion Criteria:

1. Patient refused to follow-up in our setting.
2. Patient refused to perform Trans-vaginal ultrasound in the second trimester of gestation.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: low implanted placenta women
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
The distance between lower edge of the placenta and internal os by ultrasound (millimeter) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided